CLINICAL TRIAL: NCT00395759
Title: The Visual Effect of an Investigational Artificial Tear in the Tear Layer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Collaborators: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCCO2-2233
Record Dates: First submitted 2006-11-02; First posted 2006-11-03 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2007-10

CONDITIONS: Dry Eye Disease
Keywords: contrast sensitivity
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Optiva artificial tear by Allergan

SUMMARY:
The purpose of this study is to investigate how the addition of a new artificial tear product when applied to the tear layer affects contrast sensitivity and optical aberrations over time. We will also determine if there are any adverse effects associated with drop instillation.

DETAILED DESCRIPTION:
Artificial tears are applied to the eye to treat a variety of eye conditions. These conditions typically are associated with dry eyes and include tear film deficiency due to ocular or systemic disease, lid resurfacing problems, and contact lens wear. The artificial tears are used to alleviate the dry eye symptoms. The administration of an artificial tear to the eye can disrupt the tear layer and this disruption could then result in a decrease in contrast sensitivity.1 - 6

Temporal changes in tear film structure (e.g., drying of the tear layer) can distort the optical wavefront as it passes through the tear layer and subsequently reduce contrast sensitivity.1 Theoretically, any substance applied to the tear layer that alters its structure could affect contrast sensitivity. Previous work in our lab has demonstrated that Refresh Liquigel when applied to the tear layer of non-contact and contact lens wearing subjects can decrease contrast sensitivity.4, 5, 7 In this study, we propose to examine the effects of a new investigational artificial tear on contrast sensitivity and optical aberrations for up to 30 minutes after administration into the tear layer of normal and dry eye subjects. A questionnaire will also be used to determine the opinions of the subjects concerning this new artificial tear.

ELIGIBILITY:
Inclusion Criteria:

* Thirty subjects free from ocular pathology will be chosen. Ten of the subjects will have a normal tear layer, ten will have a mild dry eye, and ten will have a moderate/severe dry eye. All subjects will be over the age of 18. Best corrected visual acuities will be at least 20/25 on a standard Snellen acuity chart at distance.

Exclusion Criteria:

* Subjects will be excluded from this project if they have, or during the course of the experiment they develop, an allergy to the eye drops used in this project.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity and optical aberrations before daily artificial tear use and at 1 and 2 weeks after daily use
Dry eye questionnaire before and at 1 and 2 weeks after artificial tear use
Slit lamp exam before and at 1 and 2 weeks after artificial tear use

CONTACTS AND LOCATIONS:
Overall Officials: William Ridder, OD. PhD, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States

REFERENCES:
- [Background] Thai LC, Tomlinson A, Ridder WH. Contact lens drying and visual performance: the vision cycle with contact lenses. Optom Vis Sci. 2002 Jun;79(6):381-8. doi: 10.1097/00006324-200206000-00012. PMID 12086305